CLINICAL TRIAL: NCT00121043
Title: An Open Label, Randomized, Crossover Study to Assess Acceptability and Functionality of SimpleJectTM Vs Pre-Filled Syringe(s) Using Kineret® (Anakinra) in Rheumatoid Arthritis (RA) Subjects Using A Self-Reported Questionnaire
Brief Title: Evaluating Kineret® (Anakinra) in Rheumatoid Arthritis (RA) Subjects Using aSelf-Reported Questionnaire
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Organization: Swedish Orphan Biovitrum (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20020125
Record Dates: First submitted 2005-06-30; First posted 2005-07-21 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Inflammation; Interleukin-1 (IL-1), r-metHuIL-1ra; Autoimmune, Kineret®; Anakinra, Immunex; Amgen, Clinical Trials
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

INTERVENTIONS:
Device: SimpleJectTM
Drug: Kineret® (Anakinra)

SUMMARY:
The primary purpose of this study is to assess the ease-of-use of SimpleJectTM compared to pre-filled syringe(s) when using Kineret® in RA subjects. The secondary purpose of this study is to assess the level of fear and anxiety associated with the use of both injection methods, to assess safety when using SimpleJectTM and to evaluate the Ease-of-Administration Questionnaire (EAQ) in terms of the quality of items, item performance, and the instrument reliability.

ELIGIBILITY:
Inclusion Criteria: - Subjects must be diagnosed with RA as guided by ACR criteria - Subjects must have an inadequate response to methotrexate alone - Subjects must receive concomitant treatment with methotrexate during the study period - Before any study specific procedure, the subject must give informed consent for participation in the study Exclusion Criteria: - Subject has previous experience using SimpleJectTM - Prior treatment with Kineret® and/or etanercept - Less than 6 weeks wash-out period for patients receiving prior infliximab treatment - Subject is currently enrolled in other clinical trial, is receiving other investigational agent(s), or at least a 30 day period has not elapsed since completion of other investigational trials with device(s) or drug(s) - Subject currently has an infection requiring systemic anti-infective therapy - Baseline neutropenia (less than 1.5 x 10^9/l) - Subjects with severe renal impairment (CLCR less than 30 ml/minute) - Subjects not willing to use adequate birth control methods - Women of childbearing potential who are pregnant, are breast-feeding or plan on becoming pregnant during the study - Planned administration of live vaccines during study period - Subject is not available for follow-up assessments - Subjects with a known sensitivity to Kineret® or any of the excipients of E. coli derived proteins - Pre-existing malignancies - Any other condition that in the investigators opinion would preclude the subject from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Difference in the EAQ Part B Ease of Use Subscale Score between the two injection methods

SECONDARY OUTCOMES:
Difference between the two injection methods for the following
EAQ Part B Total Score.
EAQ Part B Overall Satisfaction Subscale Score.
EAQ Part B Anxiety/Fear of Needles Subscale Score.
EAQ Part B Confidence in Ability of Use Subscale Score.
EAQ Part B Pain/Discomfort Subscale Score.
EAQ Part C Total Preference Score.
EAQ Quality Measures.
EAQ Item Performance Measures.
EAQ Instrument Reliability Measures.
Incidence and severity of AE's.
Incidence of concomitant medications.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com